CLINICAL TRIAL: NCT03035591
Title: Safety and Pharmacokinetics of ODM-207 in Patients With Selected Advanced Solid Tumours: an Open-label, Non-randomised, Uncontrolled, Multicentre, First-in-human Study With Cohort Expansion
Brief Title: ODM-207 in Patients With Advance Solid Tumours
Acronym: BETIDES
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Orion Corporation, Orion Pharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 3121001
Record Dates: First submitted 2017-01-20; First posted 2017-01-30 (Estimated); Last update posted 2019-10-15 (Actual); Status verified 2019-10

CONDITIONS: Solid Tumors
MeSH Terms: interventions — ODM-207

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- ODM-207 (Experimental): Escalating doses of ODM-207
  Interventions: Drug: ODM-207

INTERVENTIONS:
Drug: ODM-207

SUMMARY:
This is a first-in-man study to assess the safety and tolerability and to characterise the pharmacokinetics of ODM-207.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically or cytologically confirmed locally advanced or metastatic cancer for which no effective standard therapy exists or are refractory or resistant to conventional therapy
* Life expectancy >12 weeks
* Patient may have either measurable or non-measurable disease, but must have disease that can be evaluated for improvement of progression
* ECOG performance status of 0 to 1

Exclusion Criteria:

* History of bleeding disorder or significant bleeding episode within 6 months prior to study treatment
* Subjects receiving anticoagulants or medications that durably inhibit platelet function (7-day wash-out prior to study treatment)
* History of or current leptomeningeal or brain metastasis or spinal cord compression.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2016-12-22 (Actual); Primary Completion 2019-05-10 (Actual); Study Completion 2019-05-10 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose | 28 days
  Highest dose level at which <33% of patients in a cohort experience Dose Limiting Toxicity (DLT)

CONTACTS AND LOCATIONS:
Overall Officials: Johann De Bono, Principal Investigator — ICR/Royal Marsden
Locations (1):
- Helsinki University Central Hospital, Department of Oncology, Helsinki, Finland

REFERENCES:
- [Derived] Ameratunga M, Brana I, Bono P, Postel-Vinay S, Plummer R, Aspegren J, Korjamo T, Snapir A, de Bono JS. First-in-human Phase 1 open label study of the BET inhibitor ODM-207 in patients with selected solid tumours. Br J Cancer. 2020 Dec;123(12):1730-1736. doi: 10.1038/s41416-020-01077-z. Epub 2020 Sep 29. PMID 32989226